CLINICAL TRIAL: NCT01917825
Title: An Open-Label, Sequential, Dose Escalation Study of the Pharmacokinetics, Safety, and Preliminary Efficacy of MDT-15 in Subjects With Lumbosacral Radiculopathy
Brief Title: A Study of the Pharmacokinetics, Safety, and Preliminary Efficacy of MDT-15 in Subjects With Lumbosacral Radiculopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P12-06
Record Dates: First submitted 2013-07-30; First posted 2013-08-07 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-02

CONDITIONS: Sciatica; Lumbosacral Radiculopathy
Keywords: radicular pain
MeSH Terms: conditions — Sciatica | interventions — MDT-15 protein, C elegans

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MDT-15 (Experimental): The treatments will be administered to separate, sequential cohorts of 18 treated subjects in the following escalating doses:1 pellet, 3 pellets, and 6 pellets.
  Interventions: Drug: MDT-15

INTERVENTIONS:
Drug: MDT-15

SUMMARY:
The primary objectives of this clinical trial are to investigate the pharmacokinetics and safety of MDT-15 pellets in escalating sequential doses administered to different cohorts. Preliminary efficacy data will also be collected for assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Be male or female at least 18 years of age.
2. Have radiating pain toward the buttock down to the leg and/or feet, unilateral.
3. Have radiologic pathology change from L1 - S1 consistent with a disc protrusion, non-sequestered extrusion, or sequestered fragment, as evidenced by magnetic resonance imaging (MRI), that is consistent with the clinical signs and symptoms of lumbar radiculopathy. The MRI must have been performed within 2 months prior to screening or it will need to be repeated.
4. Have primary leg pain with an average NRS score equal to or greater than 5 as measured twice a day for five days in each of two weeks during screening.
5. Have failed conservative care for at least 6 weeks. The subject must have been treated non-operatively (e.g., bed rest, physical therapy, medications, TENS, and/or manipulation) for a period of at least 6 weeks.
6. Be willing to stop current anti-inflammatory therapy taken for treatment of radicular pain.
7. Be willing and able to keep a diary that will record study-related information.
8. If sexually active female of childbearing potential, be willing to use an acceptable method of birth control during the study. Acceptable methods include oral contraceptives (the pill), IUDs, contraceptive implants under the skin, contraceptive rings or patches or injections, diaphragms with spermicide, and condoms with spermicide. Surgical sterilization by tubal ligation or hysterectomy is acceptable. Women of child bearing potential are defined as women who are <12 months since their last menstrual cycle prior to screening and have not experienced surgical menopause.
9. Be able to understand the study and provide written informed consent.

Exclusion Criteria:

1. Have a history of lumbar surgery, including vertebroplasty and kyphoplasty.
2. Be ≤ 6 weeks after lumbar ESI or nerve block at start of screening.
3. Have current radicular pain for more than 6 months.
4. Have more than one epidural steroid injection at the affected level to be treated within the last 6 months.
5. Have demonstrated radiographic changes consistent with subject's symptoms at more than one level on the baseline MRI.
6. Have symptomatic spinal stenosis of central origin at any level based on CT myelogram or MRI.
7. Have pain that is localized in the lower back or other sites and is a greater component of the subject's total pain than the pain in the lower leg and/or foot.
8. Have physical problems that may interfere with any study assessments.
9. Have known infection with human immunodeficiency virus, hepatitis B virus, or hepatitis C virus.
10. Have presence of local or systemic malignant disease or history of local or systemic malignant disease in the past 5 years (history of basal cell carcinoma will be allowed).
11. Have impaired renal function (creatinine >1.5 times upper limit of normal).
12. Have chronic impairment liver function (aspartate aminotransferase [AST] or alanine aminotransferase [ALT] >3 times upper limit of normal).
13. Have insulin-dependent diabetes or uncontrolled diabetes mellitus (glycosylated hemoglobin [HbA1c] >7%).
14. Have leukopenia (<3,500 leukocytes/uL).
15. Have current orthostatic hypotension (defined as systolic blood pressure decrease of at least 20 mmHg or a diastolic blood pressure decrease of at least 10 mmHg or an increase in heart rate by 20 beats per minute within 3 minutes of standing).
16. Have clinically significant risk for hypotension (e.g., hypotension defined as systolic reading <90 mmHg and/or diastolic <60 mmHg, hypovolemia, autonomic neuropathy, or other medical conditions affected by changes in blood pressure).
17. Any clinically significant cardiovascular condition as evidenced by physical exam, medical history and/or baseline electrocardiogram (ECG).
18. Have evidence of bradycardia as shown by heart rate of <60 beats per minute via screening ECG.
19. Have any poorly-controlled or serious medical condition, psychiatric illness, or clinically significant laboratory value that, in the opinion of the investigator, could compromise the safety of the subject or the scientific integrity of the study (e.g., uncontrolled hypertension, autoimmune disease, or clinically relevant symptoms of thyroid dysfunction).
20. Have cauda equina syndrome.
21. Have neurological deficits, as determined by the investigator, which would interfere with the assessments required by the protocol.
22. Have been previously diagnosed with peripheral neuropathy.
23. Have vascular claudication, as determined by the investigator, which would interfere with the assessments required by the protocol.
24. Have a history or evidence of bleeding disorder (e.g., hemophilia, disseminated intravascular coagulation disorder [DIC], or thrombocytopenia [TCP])
25. Have greater than 3 mm spondylolisthesis at the affected level.
26. Have BMI greater than or equal to 40, or with any anatomic issues that may interfere with placement of the MDT-15 pellets as noted by the Investigator.
27. Have a diagnosis of major depression.
28. Have sustained a vertebral or hip fracture within the last year.
29. Have known or suspected allergy or hypersensitivity to clonidine, lidocaine, contrast media, opioids, any medication that may be given as part of the site's standard of care related to the study drug implantation procedure, or any other medication that may be given as treatment during the study.
30. Have a known or suspected allergy to polylactic acid (found in products such as Lupron Depot®, Atridox®, some types of dermal fillers, and some types of sutures).
31. If female, be pregnant or breastfeeding, or desiring to become pregnant during the trial.
32. Have taken an investigational drug or used an investigational device within the past 30 days or intending to use an investigational drug or device during the trial.
33. Have active alcoholism or drug dependency, as determined by the investigator
34. Be currently on worker's compensation or in litigation related to injury or medical condition.
35. Be in circumstances which make it difficult to maintain a usual nighttime sleep schedule (e.g., the subject works on an evening/night shift or otherwise has a work or activity schedule which could confound or interfere with study assessments).
36. Have current treatment with any of the following medications:

    1. Systemic corticosteroids (intranasal/inhaled steroids are acceptable).
    2. Immunosuppressant therapy to treat autoimmune diseases (e.g., rheumatoid arthritis, multiple sclerosis, myasthenia gravis, systemic lupus erythematosus, sarcoidosis, focal segmental glomerulosclerosis, Crohn's disease, Behcet's Disease, pemphigus, and ulcerative colitis).
    3. Oral or topical products that contain clonidine (e.g., Catapres).
    4. Herbal supplements that contain yohimbine.
    5. Anti-coagulant therapy (prophylactic aspirin at 81mg/day is acceptable). If applicable, aspirin therapy should be held before and after the study procedure based on the investigator's discretion.
    6. Calcium channel blocker, digoxin, or beta-adrenergic blockers.
37. Have chronic use of opioids (including tramadol), defined as use 20 out of the last 30 days prior to study screening.
38. Have emotional or health concerns (in the judgment of the investigator) that may compromise the safety of the subject, may make compliance difficult, or may confound the reliability of information acquired in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-07; Primary Completion 2015-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Cmax | 84 days
  The Pharmacokinetics profile (Cmax, Tmax, AUC0-t, and AUC0-∞) following administration of up to six MDT-15 pellets in escalating sequential doses to different cohorts will be evaluated.
Tmax | 84 days
  The Pharmacokinetics profile (Cmax, Tmax, AUC0-t, and AUC0-∞) following administration of up to six MDT-15 pellets in escalating sequential doses to different cohorts will be evaluated.
AUC0-t | 84 days
  The Pharmacokinetics profile (Cmax, Tmax, AUC0-t, and AUC0-∞) following administration of up to six MDT-15 pellets in escalating sequential doses to different cohorts will be evaluated.
AUC0-∞ | 84 days
  The Pharmacokinetics profile (Cmax, Tmax, AUC0-t, and AUC0-∞) following administration of up to six MDT-15 pellets in escalating sequential doses to different cohorts will be evaluated.
Incidence of Adverse Events | 364 days
  Incidence of Adverse Events as a Measure of Safety.

SECONDARY OUTCOMES:
Change in Radicular Leg Pain | Baseline and 364 days
  Radicular leg pain measured by a 0-10 Numeric Rating Scale (NRS).
Change in Physical Function | Baseline and 364 days
  Physical Functioning measured by the Modified Roland Disability Questionnaire (RMS-L).
Change in Back Pain | Baseline and 364 days
  Back pain measured by a 0-10 Numeric Rating Scale (NRS).
Change in Neuropathic Type Symptoms | Baseline and 84 days
  Neuropathic Type Symptoms as measured by the Short-form McGill Pain Questionnaire (SF-MPQ-2).
Change in Medical Outcomes study - Sleep Scale | Baseline and 84 days
  Sleep as measured by the Medical Outcomes Study - Sleep Scale (MOS-Sleep).
Change in Emotional Function | Baseline and 84 days
  Emotional functioning as measured by the Profile of Mood States - Brief Form (POMS- Brief).
Change in Work Function | Baseline and 84 days
  Work Function as measured by the Work Limitations Questionnaire (WLQ).
Global Rating of Improvement | 84 days
  Global rating of improvement as measured by a Patient Global Impression of Change (PGIC).

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Holy Cross Orthopedic Institute, Fort Lauderdale, Florida
  - Millennium Pain Center, Bloomington, Illinois
  - Indiana Spine Group, Carmel, Indiana
  - Franciscan St Francis Pain and Spine Center, Indianapolis, Indiana
  - Otrimed Clinical Research, Edgewood, Kentucky
  - Pain and Rehabilitation Specialists, St Louis, Missouri